## **COVER PAGE (IDENTIFYING INFORMATION)**

#### Official Title:

The Longitudinal Impact of Prenatal Pilates on Female Sexual Function and Sexual Distress During Pregnancy

## **Protocol Record ID (Local):**

OKAN-PP-FSFI-2025

### **ClinicalTrials.gov Identifier:**

NCT number not yet assigned (pending registration)

## **Document Type:**

Informed Consent Form

### **Document Date / Version:**

Version 1.0 – 04 Feb 2026

# **Sponsor / Institution:**

Istanbul Okan University Hospital, Department of Obstetrics and Gynecology

#### INFORMED CONSENT FORM

## **Study Title**

The Longitudinal Impact of Prenatal Pilates on Female Sexual Function and Sexual Distress During Pregnancy

## **Invitation to Participate**

You are invited to take part in a research study conducted at **Istanbul Okan University Hospital, Department of Obstetrics and Gynecology**. Before you decide whether to participate, please read the information below carefully. You may ask any questions at any time.

## **Purpose of the Study**

The purpose of this study is to compare **female sexual function (FSFI)** and **sexual distress (FSDS-R)** between pregnant women who regularly practice **prenatal Pilates** and those who do not.

This study is an **observational study**. No exercise program will be prescribed or assigned by the research team. Data will be collected only through questionnaires.

## **Study Procedures**

If you agree to participate, you will be asked to complete questionnaire forms during pregnancy.

No medical procedures will be performed as part of this study.

No blood or tissue samples will be taken, and no additional tests will be required.

## **Voluntary Participation and Withdrawal**

Participation in this study is entirely voluntary. You may refuse to participate or withdraw from the study at any time, with or without giving a reason, and without any effect on your medical care.

#### **Benefits**

You may not receive any direct benefit from participating in this study. However, the results may help improve understanding of the effects of physical activity on sexual health during pregnancy and may contribute to future counseling and supportive care for pregnant women.

#### **Risks and Discomforts**

There are no expected physical risks because no medical procedures will be performed. Some questions may be personal or sensitive and may cause mild emotional discomfort. You may skip any question you do not wish to answer.

## Confidentiality

All information collected during this study will be kept confidential. Your personal identity will not appear in any study records, reports, or publications. Data will be anonymized and used only for scientific purposes.

## **New Information**

If new information becomes available that may affect your willingness to continue participating, you will be informed in a timely manner. If any condition arises that requires termination of your participation, you will also be informed.

### **Contact Information**

If you have any questions or concerns about this study or your participation, you may contact the research team at any time:

Principal Investigator: Gökçenur Karakelleoğlu, MD

**Phone:** +90 532 670 2049

Study Site Address: İçmeler Mah. Aydınlı Cad. No: 2, Istanbul Okan University Hospital, Tuzla,

Istanbul, Turkey

### **Consent Statement**

Participant (Volunteer)

I confirm that I have received written and verbal information about the research study described above from the physician/researcher whose name is written below. I understand that my participation is voluntary and that I may withdraw from the study at any time, with or without a reason.

By signing below, I agree to participate in this study voluntarily, without any pressure or influence.

| . a | |
|--------------|---------------------------------|
| Full Name: _ | |
| Date: / | / |
| Signature: | |
| Physician/Re | esearcher Providing Information |
| Full Name: _ | |
| Date:/ | / |
| Signature: | |